CLINICAL TRIAL: NCT06959914
Title: The Effect of Arteriovenous Fistula Care Training Given to Hemodialysis Patients on Quality of Life, Comfort and Self-Care Behaviours
Acronym: Fistula care
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kafkas University (Other)
Responsible Party: Principal Investigator, Zümrüt AKGÜN ŞAHİN, Assoc.Prof, Kafkas University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 0000-0001-7141-273X
Record Dates: First submitted 2025-04-21; First posted 2025-05-07 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-05

CONDITIONS: Hemodialysis Patient; Hemodialysis Catheter
Keywords: Arteriovenous Fistula; Qualitiy of life; Comfort; Self-care; Hemodialysis; Hemodialysis access
MeSH Terms: conditions — Arteriovenous Fistula | interventions — Sensitivity Training Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Control group (Active Comparator): HD patients who fulfil the inclusion criteria will be met face-to-face. Patients who agree to participate in the study will be asked to sign an informed consent form. Afterwards, Patient Information Form, SF-12 Quality of Life Short Form, Comfort Scale for Hemodialysis Patients and Scale for Evaluation of Self-Care Behaviours Regarding Arteriovenous Fistula in Hemodialysis Patients will be given to the patients and those who can read and write will be asked to fill them in by themselves. For illiterate patients, pre-test data will be collected by reading the questionnaire forms by the investigators. No treatment will be applied to the participants in this group. At the end of 8 weeks, all participants will be asked to fill in the Patient Information Form, SF-12 Quality of Life Short Form, Comfort Scale for Hemodialysis Patients and Self-Care Behaviour Assessment Scale for Arteriovenous Fistula in Hemodialysis Patients as a post-test application.
  Interventions: Other: Training group

INTERVENTIONS:
Other: Training group — Patients in the intervention group will receive AVF care training. The training will last for 8 weeks and is planned to be given once a week. In the first session, the patients in the intervention group will be introduced. Afterwards, general information will be provided about the purpose and applications of AVF training and the importance of participation in training will be emphasized. Afterwards, patients who agree to participate in the study will sign an informed consent form. In addition, the Patient Information Form, SF-12 Quality of Life Short Form, the Comfort Scale for Hemodialysis Patients and the Scale for Assessing Self-Care Behaviors Related to Arteriovenous Fistula in Hemodialysis Patients will be given and asked to answer. For those who cannot read or write, the researchers will read the survey forms. In the first session, the pre-test data of the patients will be collected and then the training books will be given.

SUMMARY:
This study will be conducted to evaluate the effect of Arterio-Venous Fistula (AVF) care training given to hamodialysis patients on quality of life, comfort and self-care behaviours. Patient education is one of the practices that help patients to gain self-care behaviours as well as reducing the cost of health expenditures. Nurses are health professionals who play an important role in patient education. Nurses provide patient education by using different materials. These materials can sometimes be mobile phones, videos, web-based applications, sometimes face-to-face interviews with patients, brochures or written materials. In this study, a training programme for AVF care will be developed. In addition, it is expected that the AVF care training to be given to HD patients will increase the quality of life and comfort areas, and increase the awareness and well-being levels of patients in self-care behaviours. The effectiveness of the study will be expanded by presenting the results of the research as a paper in an international comprehensive congress. An article of the study will be published in a journal scanned in international indexes and will be included in the literature.

DETAILED DESCRIPTION:
This study will be conducted to determine the effect of Arterio-Venous Fistula (AVF) care training given to haemodialysis patients on quality of life, comfort and self-care behaviours.

The research will be conducted as an experimental, pre-test post-test randomised controlled experimental study.

Hypotheses:

H0: AVF care training given to haemodialysis patients has no effect on patients' quality of life, comfort and self-care behaviours.

H1: AVF care training given to haemodialysis patients affects patients' quality of life.

H2: AVF care training given to haemodialysis patients affects patients' comfort.

H3: AVF care training given to haemodialysis patients affects patients' self-care behaviours.

The research population will consist of a total of 67 patients receiving HD treatment in the Dialysis Unit and having AVF. Similar study data were taken into consideration in the selection of the research sample. As a result of the power analysis performed in the G*Power version 3.1.9.7 programme, it was determined that a total of 52 participants, at least one person for each of the intervention and control groups, should be included in the sample size, 95% confidence interval, 95% test power (1-ß), 0.05% margin of error level.

Randomisation and Blinding Simple random sampling method will be used for randomisation of the study. In order to avoid interactions between the patients participating in the study, they will be grouped according to the days of HD treatment sessions. In Group I: Patients receiving HD treatment on Mondays, Wednesdays and Fridays, and in Group II; patients receiving HD treatment on Tuesdays, Thursdays and Saturdays. Which group will be the control group and which will be the intervention group will be decided by drawing lots.

Inclusion Criteria for the Study:

* Volunteering to participate in the study,
* Speak Turkish.
* Being 18 years old and above
* Having an AVF
* Being on the floor for HD at least 3 times in 6 weeks
* Not having treatments or mental problems that prevent participation in the study

Exclusion Criteria for the Study:

* Not consenting to participate in the study
* Having a diagnosed psychiatric illness,
* Having a visual, hearing, speech, physical or mental disability,
* Dropping out of education. Data Collection Tools Data will be collected using the "Patient Information Form", "SF-12 Quality of Life Short Form ", "Comfort Scale for Hemodialysis Patients" and "Self-Care Behavior Assessment Scale for Arteriovenous Fistula in Hemodialysis Patients".

Data Collection / Intervention Procedure First, patients will be informed about the study and will be asked to sign an informed consent form. Then, all participants will fill out the questionnaire forms as a pre-test application.

No training will be given to the patients in the control group and the questionnaire forms will be applied again after 8 weeks. The patients in the intervention group will be given 8 weeks of AVF care training. At the end of the training, the questionnaire forms will be applied to the patients again and the effectiveness of the training will be evaluated.

Training Booklet Content The training booklet will be prepared using literature reviews, research results, and evidence-based practice guides. After the training booklet is created, it will be sent for expert opinion. The training booklet will include topics on fluid control, diet, and medication management.

Training Program Goals

* Knowing the functions of the kidneys
* Knowing the treatment options for chronic renal failure
* Knowing the vascular access routes used in hemodialysis
* Knowing arteriovenous fistula care
* Knowing the medications frequently used
* Knowing the meanings of laboratory findings
* Knowing the problems frequently encountered and solution suggestions

ELIGIBILITY:
Inclusion Criteria:

* -Volunteering to participate in the research,
* Speaking Turkish.
* 18 years of age or older
* Having AVF
* Receiving HD treatment 3 times a week for at least 6 months
* Not having cognitive and mental problems that prevent participation in the study

Exclusion Criteria:

* Not consenting to participate in the study

  * Being a diagnosed psychiatric individual,
  * Having a visual, hearing, speech, physical or mental disability,
  * Being incomplete in their education.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Evaluation of Self-Care Behaviours Regarding Arteriovenous Fistula in Hemodialysis Patients | eight weeks
  The scale was developed by Sousa et al. to evaluate patients' care behaviors related to arteriovenous fistula and to follow up patients' education. The scale was developed in Portuguese and its validity and reliability for the Turkish society was performed by İkiz and Usta. It is a 16-item, 5-point Likert scale consisting of single-sentence phrases. The scale consists of two sub-dimensions as symptom and "Symptom Management" and "Prevention of Complications". The item numbers of the Symptom and Symptom Management sub-dimension of the scale are 1,3,6,11,13,16 and the item numbers of the Complication Prevention sub-dimension are 2,4,5,7,8,9,10,12,14,15.22. The time required to administer the scale is about 2-3 minutes. While 16 indicates the lowest possible score in the scoring of the scale, 80 indicates the highest score. The lowest possible score from the symptom and symptom management sub-dimension is 6 and the highest score is 30. The lowest score that can be obtained from the sub-d
Comfort Scale for Haemodialysis Patients (HCP) | eight weeks
  It was revised by Orak et al. (2017) by using the General Comfort Scale developed by Kolcaba (1992) and later comfort scales developed specifically for certain situations. The scale consists of 9 items and 2 sub-dimensions (overcoming and relaxing). The responses given to the 4th item of the 5-point Likert-type scale are scored as "never" 1 point, "very rarely" 2 points, "sometimes" 3 points, "very often" 4 points and "always" 5 points. The scores given to the other items (1-3, 5-9) are scored in reverse: "never" 5 points, "very rarely" 4 points, "sometimes" 3 points, "very often" 2 points and "always" 1 point. The evaluation of the scale is determined by calculating the average score, the lowest score that can be obtained from the scale is 1, the highest score is 5. The comfort level increases as the score gets closer to 5. The scale has two sub-dimensions: "Relaxation" (items 7-9) and "Overcoming" (items 1-6).
SF-12 Quality of Life Short Form | eight weeks
  SF-12 was developed by Ware et al. (1996). The Turkish version of the scale was developed by Soylu and Kütük. The scale is an outcome measure filled out by the patient, evaluating the impact of health on the individual's daily life. SF-12 is basically a shortened version of SF36, consisting of 8 sub-dimensions and a total of 12 items. This scale evaluates physical functioning with 2 items, physical role with 2 items, body pain with 1 item, general health with 1 item, energy with 1 item, social functioning with 1 item, emotional role with 2 items, and mental health with 2 items.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sousa CN, Apostolo JL, Figueiredo MH, Dias VF, Teles P, Martins MM. Construction and validation of a scale of assessment of self-care behaviors with arteriovenous fistula in hemodialysis. Hemodial Int. 2015 Apr;19(2):306-13. doi: 10.1111/hdi.12249. Epub 2014 Dec 5. PMID 25477007
- [Background] Kang H. Sample size determination and power analysis using the G*Power software. J Educ Eval Health Prof. 2021;18:17. doi: 10.3352/jeehp.2021.18.17. Epub 2021 Jul 30. PMID 34325496
- [Background] Dilbilir Y, Kavurmaci M. Determining the effect of arteriovenous fistula care training on the self-care behaviors of hemodialysis patients. Ther Apher Dial. 2024 Dec;28(6):893-903. doi: 10.1111/1744-9987.14174. Epub 2024 Jun 13. PMID 38872366
- [Background] Wang J, Yue P, Huang J, Xie X, Ling Y, Jia L, Xiong Y, Sun F. Nursing Intervention on the Compliance of Hemodialysis Patients with End-Stage Renal Disease: A Meta-Analysis. Blood Purif. 2018;45(1-3):102-109. doi: 10.1159/000484924. Epub 2017 Dec 12. PMID 29241195
- [Background] Ramezani T, Sharifirad G, Rajati F, Rajati M, Mohebi S. Effect of educational intervention on promoting self-care in hemodialysis patients: Applying the self-efficacy theory. J Educ Health Promot. 2019 Mar 14;8:65. doi: 10.4103/jehp.jehp_148_18. eCollection 2019. PMID 31008132
- [Background] Casey JR, Hanson CS, Winkelmayer WC, Craig JC, Palmer S, Strippoli GF, Tong A. Patients' perspectives on hemodialysis vascular access: a systematic review of qualitative studies. Am J Kidney Dis. 2014 Dec;64(6):937-53. doi: 10.1053/j.ajkd.2014.06.024. Epub 2014 Aug 10. PMID 25115617
- [Background] Shamasneh AO, Atieh AS, Gharaibeh KA, Hamadah A. Perceived barriers and attitudes toward arteriovenous fistula creation and use in hemodialysis patients in Palestine. Ren Fail. 2020 Nov;42(1):343-349. doi: 10.1080/0886022X.2020.1748650. PMID 32338112
- [Background] Al-Balas A, Shariff S, Lee T, Young C, Allon M. Clinical Outcomes and Economic Impact of Starting Hemodialysis with a Catheter after Predialysis Arteriovenous Fistula Creation. Am J Nephrol. 2019;50(3):221-227. doi: 10.1159/000502050. Epub 2019 Aug 8. PMID 31394548